CLINICAL TRIAL: NCT06401785
Title: To Evaluate the Efficacy of Oral Molecular Hydrogen Supplement in Patients With Chronic Diseases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HoHo Biotech (Industry)
Collaborators: Taoyuan Armed Forces General Hospital (Unknown); Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: C202305150
Record Dates: First submitted 2024-02-18; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Chronic Disease; Chronic Inflammation
Keywords: Hydrogen supplement; Oral hydrogen capsules
MeSH Terms: conditions — Chronic Disease | interventions — Hydrogen

STUDY DESIGN:
Intervention Model Description: In experiment group, participants will receive 2 solid hydrogen capsules every day for 24 weeks. In control group, participants will receive 2 capsules not containing hydrogen every day for 24 weeks.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen capsules (Experimental): Hydrogen supplement
  Interventions: Dietary Supplement: Hydrogen capsules
- Placebo (Placebo Comparator): Placebo supplement
  Interventions: Dietary Supplement: Hydrogen capsules

INTERVENTIONS:
Dietary Supplement: Hydrogen capsules — In experiment group, participants will receive 2 solid hydrogen capsules every day for 24 weeks. In control group, participants will receive 2 capsules not containing hydrogen every day for 24 weeks.

SUMMARY:
The supplementation of hydrogen molecules as an aid, adjuvant, may speed up recovering the course of the disease. The purpose of this study is to determine the possible efficacy and safety of solid hydrogen supplements for a clinical study in patients with chronic diseases. Patients will receive hydrogen capsules with their conventional treatment for 24 weeks. Investigators will test for any changes in haematologic, urine analysis and health status during and following the exposure period.

DETAILED DESCRIPTION:
Hydrogen supplement has been shown to have significant removing effects on free radicals. International clinical trials have shown promise that hydrogen molecules may reduce chronic inflammatory and then speed up recovering the course of the disease.The purpose of this study is to determine the possible efficacy and safety of hydrogen supplements in different formula and dose exposures for a clinical study in patients with chronic diseases.Study design: 60 chronic diseases patients will be recruited from the Taoyuan Armed Forces General Hospital and Tri-Service General Hospital for this study. Participants will be screened by doctors for their eligibility and undergo a series of tests (questionnaires and examinations).Consenting participants will then be randomly allocated into 2 groups (experiment group and control group, single-blind study). In experiment group, participants will receive 2 solid hydrogen capsules every day for 24 weeks. In control group, participants will receive 2 capsules not containing hydrogen every day for 24 weeks. Participants will be examined their regular haematology, urine and health status before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 80
* Able to compliant with the protocol
* Able to return to the hospital regularly
* Patients with chronic inflammation, including patients with autoimmune diseases, metabolic-related diseases, chronic kidney disease or nephritis, tumor patients, etc.

Exclusion Criteria:

* Pregnancy
* Expected pregnancy
* Attending other clinical trials with 6 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-11 (Estimated); Primary Completion 2024-12-29 (Estimated); Study Completion 2025-01-29 (Estimated)

PRIMARY OUTCOMES:
Improvement in Blood Routine | Change from Baseline of Blood Routine, and every return per 4 weeks during 24 weeks of the intervention
  Change in Blood Routine, including WBC, RBC, HGB, HCT, MCV, MCH, MCHC, PLT, Lymphocyte, Monocyte, Eosinophil, Basophil, Neutrophil, Triglyceride, Cholesterol, HDL, LDL, ESR, and CRP
Improvement in Urine Routine | Change from Baseline of Urine Routine, and every return per 4 weeks during 24 weeks of the intervention
  Change in Urine Routine, including GLU, PRO, BIL, URO, PH, SG, OB, KET, NIT, Uric acid, BUN, and eGFR
Improvement in the Health Assessment Questionnaire Disability Index (HAQ-DI) Questionnaire | Change from Baseline of HAQ-DI, and every return per 4 weeks during 24 weeks of the intervention
  Change in the (HAQ-DI) Questionnaire
Improvement in the Disease Activity Score (DAS 28) | Change from Baseline of DAS 28, and every return per 4 weeks during 24 weeks of the intervention
  Change in the DAS 28
Improvement in the Brief Fatigue Inventory-Taiwan (BFI-T) | Change from Baseline of BFI-T, and every return per 4 weeks during 24 weeks of the intervention
  Change in the BFI-T

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Tri-Service General Hospital, Taipei
  - Taoyuan Armed Forces General Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided